CLINICAL TRIAL: NCT04416698
Title: Helping Youth to Quit Smoking by Understanding Their Risk Perception, Behaviour, and Attitudes Related to Electronic Cigarettes and Other New Tobacco Products
Brief Title: Understanding Risk Perception, Behaviour, and Attitudes Related to Other New Tobacco Products Among Youth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: other tobacco products
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Smoking Cessation
Keywords: Youth smokers smoking cessation, tobacco products
MeSH Terms: conditions — Smoking Cessation | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth smokers: Participants of Youth Quitline
  Interventions: Behavioral: Individual qualitative interview; Behavioral: cross-sectional survey study

INTERVENTIONS:
Behavioral: Individual qualitative interview — Individual interviews will be conducted to understanding the needs and concerns of youth smokers of e-cigarette or other new tobacco products, including their risk perceptions, and the behaviour, attitudes, and experiences related to these tobacco products.
Behavioral: cross-sectional survey study — structured questionnaire will be constructed for a cross-sectional survey to further explore the behaviour, attitudes, and experiences related to electronic cigarettes or other new tobacco products among youth.

SUMMARY:
To understand the risk perception, behaviour, and attitudes related to electronic cigarettes and other tobacco products among youth.

DETAILED DESCRIPTION:
Phase I Individual qualitative interviews will be conducted to understanding the needs and concerns of youth smokers of e-cigarette or other new tobacco products, including their risk perceptions, and the behaviour, attitudes, and experiences related to these products.

Phase II The findings from the interview in phase I will guide the development of a structure questionnaire for a cross-sectional survey to further explore the behaviour, attitudes, and experiences related to e-cigarette or other new tobacco products among youth.

The findings of this study have important implications for research and clinical practice. Understanding how youth smokers perceive the risks of using e-cigarette and other new tobacco products, and their behaviour, attitudes, experiences related to smoking to help them achieve smoking abstinence. Moreover, the results of this study can understand the misconceptions about e-cigarette and other new tobacco product among youth, increase their perception of the risks of continued smoking and benefits of quitting.

ELIGIBILITY:
Inclusion Criteria:

* Youth smokers who contacted the Youth Quitline will be eligible to be included in this study if they (1) are ethnic Chinese; (2) are aged ≤ 25 years; (3) are ever user of e-cigarette or any new tobacco products; and (4) spoke Cantonese.

Exclusion Criteria:

* psychologically or physically unable to communicate

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth smokers
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Smoking behaviors in phase I | Baseline
  the behaviour, attitudes, and experiences related to electronic cigarettes and other new tobacco products among youth in individual qualitative interview (Phase I)
Smoking behaviors in phase II | Baseline
  the behaviour, attitudes, and experiences related to electronic cigarettes and other new tobacco products among youth in structured questionnaires (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Pokfulam, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)